CLINICAL TRIAL: NCT05931133
Title: Urdu Translation and Validation of Michigan Hand Outcome Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/0029 Alishfa zahoor
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Upper Extremity Problem
Keywords: URDU VERSION, MICHIGAN HAND OUTCOME QUESTIONAIRE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NO INTERVENTION — NO INTERVENTION WILL BE GIVEN

SUMMARY:
Aim of this study to provide a urdu version of Michigan Hand Outcome Questionnaire, that will be more understandable for Pakistani People.

DETAILED DESCRIPTION:
Because of these unique qualities, the MHQ has become one of widely used tools by the clinicians to assess quality-of-life relevant to functioning of hands and upper limb. It has also been translated to many other languages from the original English version for an easy understanding and adaptation into the local population. despite being its availability in approximately 20 different languages., the Urdu translation of this questionnaire has not yet been published anywhere. Urdu is Pakistan's official language, and the majority of Pakistanis are unable to understand this subjective assessment questionnaire originally written in English. It is required to translate the questionnaire into Urdu for Pakistanis people as the upper limb disorders are one of the most prevalent musculoskeletal disorders in Pakistan. Urdu translation of Michigan Hand Outcomes Questionnaire will help the Pakistan population with hand disorders to describe their pain or disability experience clearly. The Clinical physiotherapists of Pakistan can be capable of capturing the subjective health states of Pakistani patients with hand disorders more conveniently using the Urdu translated MHQ.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with conditions and diseases of the Hand and the Upper extremity (arthritis, trauma etc.).

  * Both genders of age 18 and over
  * Patients who are willing to fill study questionnaires.

Exclusion Criteria:

* • Unable to read or write in Urdu

  * People with cognitive dysfunction
  * People with Any neurological disorder
  * Unable to fill questionnaire independently

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the participants with upper limb and hand disorders will be required to fill the urdu version of michigan hand outcome questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Each question of Urdu version of Michigan hand outcome questionnaire | 6-8 weeks
  AS its a validity and reliability study so each question of questionnaire will be outcome

SECONDARY OUTCOMES:
Each question of Urdu version of SF-36 questionnaire | 6-8 Weeks
  AS its a validity and reliability study so each question of questionnaire will be outcome

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, Masters, Principal Investigator — Riphah International University
Locations (1):
- District Health quarter jhang, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung KC, Pillsbury MS, Walters MR, Hayward RA. Reliability and validity testing of the Michigan Hand Outcomes Questionnaire. J Hand Surg Am. 1998 Jul;23(4):575-87. doi: 10.1016/S0363-5023(98)80042-7. PMID 9708370
- [Background] Chung KC, Hamill JB, Walters MR, Hayward RA. The Michigan Hand Outcomes Questionnaire (MHQ): assessment of responsiveness to clinical change. Ann Plast Surg. 1999 Jun;42(6):619-22. doi: 10.1097/00000637-199906000-00006. PMID 10382797
- [Background] Blomstrand J, Karlsson J, Fagevik Olsen M, Kjellby Wendt G. The Michigan Hand Outcomes Questionnaire (MHQ-Swe) in patients with distal radius fractures-cross-cultural adaptation to Swedish, validation and reliability. J Orthop Surg Res. 2021 Jul 7;16(1):442. doi: 10.1186/s13018-021-02571-7. PMID 34233700